CLINICAL TRIAL: NCT01654640
Title: Phase 4 Study of Metformin on Obesity and Metabolic Disturbance in Patients Taking Clozapine
Brief Title: The Effect of Metformin on Obesity and Metabolic Disturbance in Patients Taking Clozapine
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Failure to recruit the planned number of participants
Sponsor: Seoul National University Hospital (Other)
Collaborators: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Principal Investigator, Yong Min Ahn, professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DW_Metformin
Record Dates: First submitted 2012-07-16; First posted 2012-08-01 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Schizophrenia
Keywords: schizophrenia; obesity; clozapine; metformin
MeSH Terms: conditions — Schizophrenia; Obesity | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin group (Experimental): Metformin 500mg 1 tablet p.o. bid
  Interventions: Drug: Metformin
- Placebo group (Placebo Comparator): 1 tablet p.o. bid
  Interventions: Drug: Placebo (for metformin)

INTERVENTIONS:
Drug: Metformin — metformin 500mg p.o. bid for 24 weeks
  Other Names: Diabex
  Arms: Metformin group
Drug: Placebo (for metformin) — placebo 1T bid
  Other Names: placebo
  Arms: Placebo group

SUMMARY:
The purpose of this study is the evaluation of effect of metformin on obesity and metabolic disturbance in patients taking clozapine.

DETAILED DESCRIPTION:
In this study, the investigators are going to examine the effect of metformin on obesity and metabolic disturbance in patients with schizophrenia who have taken clozapine.The metformin 500mg will be administrated per oral twice a day for 24 weeks and for control group, placebo will be given same route and process.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 ~ 65
* Patient with schizophrenia according to DSM-IV criteria
* Patient have signed on the informed consent, and well understood the objective and procedure of this study.
* Patient taking clozapine 3months or more
* Patient increased in weight more than 10 % of that of before antipsychotics use

Exclusion Criteria:

* Patient taking other antipsychotics with clozapine
* Patient in treatment of diabetes
* Patient in treatment of dyslipidemia
* Allergy or hypersensitivity to metformin
* Pregnant or breast-feeding female patient.
* Patient with severe medical condition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
change of weight | baseline, 12 weeks, 24 weeks
  change of weight after 12-week, 24-week. calculation; (weight of 12-week - weight of baseline)/baseline weight (weight of 24-week - weight of baseline)/baseline weight

SECONDARY OUTCOMES:
Positive and Negative Symptom Scale(PANSS) | baseline, 12 weeks, 24 weeks
  baseline, 1-week, 4-week, 12-week, 24-week(end-point)
MADRS(montgomery asberg depression rating scale) | baseline, 12 weeks, 24 weeks
  baseline, 1-week, 4-week, 12-week, 24-week(end-point)
Clinical Global Impression-severity(CGI-S) | baseline, 6 weeks, 24 weeks
  baseline, 1-week, 4-week, 12-week, 24-week(end-point)
Clinical Global Impression-improvement(CGI-I) | baseline, 12 weeks, 24 weeks
  baseline, 1-week, 4-week, 12-week, 24-week(end-point)
Beck's Depression Inventory(BDI) | baseline, 12 weeks, 24 weeks
  baseline, 1-week, 4-week, 12-week, 24-week(end-point)
Liverpool University Neuroleptic Side Effect Rating Scale(LUNSERS) | baseline, 12 weeks, 24 weeks
  baseline, 1-week, 4-week, 12-week, 24-week(end-point)
World Health Organization Quality of Life-BREF (WHOQOL-BREF) | baseline, 12 weeks, 24 weeks
  baseline, 1-week, 4-week, 12-week, 24-week(end-point)
Short form(36) Health survey (SF-36) | baseline, 12 weeks, 24 weeks
  baseline, 1-week, 4-week, 12-week, 24-week(end-point)
abdominal fat amount CT | baseline, 12 weeks, 24 weeks
  baseline, 12-week, 24-week
change of prevalence of metabolic syndrome | baseline, 12 weeks, 24 weeks
  waist circumference, blood pressure cholesterol,triglyceride, HDL-cholesterol,fasting glucose

CONTACTS AND LOCATIONS:
Overall Officials: Yong Min Ahn, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- See also: study site — http://www.snuh.org/